CLINICAL TRIAL: NCT05901285
Title: Phase 1 Study of Intratumoral Administration of VAX014 With Expansion in Combination With a Checkpoint Inhibitor in Subjects With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vaxiion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VX0120
Record Dates: First submitted 2023-05-24; First posted 2023-06-13 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumor; Advanced Solid Tumors Appropriate for Treatment With Either Nivolumab or Pembrolizumab
MeSH Terms: interventions — Nivolumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VAX014 (Dose Escalation) (Experimental): Dose escalation of VAX014 [recombinant bacterial minicells (rBMCs)] intratumoral injections alone for subjects with solid tumors relapsed and/or refractory to standard treatment and appropriate for injection of a nodal, subcutaneous, or cutaneous tumor via palpation or with the assistance of ultrasound.
  Interventions: Drug: VAX014
- VAX014 in Combination with Either Nivolumab or Pembrolizumab (Dose Expansion) (Experimental): Dose expansion of VAX014 [recombinant bacterial minicells (rBMCs)] intratumoral injections in combination with Investigator's choice of nivolumb or pembrolizumab for subjects with solid tumors relapsed and/or refractory to standard treatment and appropriate for injection of a nodal, subcutaneous, or cutaneous tumor via palpation, with the assistance of ultrasound, or interventional radiology.
  Interventions: Drug: VAX014; Combination Product: Nivolumab or pembrolizumab

INTERVENTIONS:
Drug: VAX014 — Intratumorally administered oncolytic agent comprised of recombinant bacterial minicells. VAX014 is not infectious and is not capable of replication
Combination Product: Nivolumab or pembrolizumab — VAX014 will be given in combination with Investigator's choice of nivolumab or pembrolizumab.
  Arms: VAX014 in Combination with Either Nivolumab or Pembrolizumab (Dose Expansion)

SUMMARY:
The purpose of this research study is to evaluate the safety, tolerability and activity of VAX014 for intratumoral injections (VAX014) as a single agent as well as in combination with Investigator's choice of nivolumab or pembrolizumab in patients with advanced solid tumors. VAX014 is a targeted oncolytic agent designed to kill tumor cells following intratumoral injection into advanced solid tumors.

DETAILED DESCRIPTION:
This study will evaluate the safety and tolerability of VAX014 using a 3+3 dose escalation design to determine a maximum tolerated dose (MTD) or maximum practical dose (MPD) of single agent VAX014. The DLT assessment period will be the initial 21-days of injections. Subjects will receive weekly injections for the initial 8 weeks. Up to six dose levels will be evaluated (i.e., [starting dose], [starting dose] x 3, [starting dose] x 10, [starting dose] x 30, [starting dose] x 100, [starting dose] x 300).

Subjects may continue on treatment following discussion between the Principal Investigator and Sponsor/Medical Monitor.

After the determination of a single agent RP2D by the SRC for single agent intratumoral VAX014, an Expansion Phase will be conducted combining intratumoral VAX014 with Investigator's choice of nivolumab or pembrolizumab. The SRC may adjust the RP2D of VAX014 used during the Expansion Phase based on accumulating safety data.

The Expansion Phase will consist of up to 25 subjects. For the first 3 subjects treated with the combination of VAX014 and either nivolumab or pembrolizumab, the initial 2 doses of intratumoral VAX014 will be reduced by one dose level from the VAX014 RP2D. If the initial 3 subjects are able to escalate to the RP2D for VAX014, all subsequent subjects will then receive VAX014 at the RP2D starting with the first dose of VAX014.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18+
2. Informed consent
3. Histological or cytopathological confirmed diagnosis of a locally advanced or metastatic solid tumor
4. Progression following at least one prior standard treatment or intolerant of standard treatments.
5. [Dose Escalation] Availability of archival or fresh tumor tissue
6. [Expansion] Willing to undergo biopsy of the tumor to be injected prior to the initial VAX014 injection (may provide archival tissue instead if approved by Medical Monitor)
7. No available SOC therapy that would confer clinical benefit
8. [Dose escalation] At least one cutaneous, subcutaneous, or nodal injectable tumor (between 1 and 10 cm in largest diameter) that can be injected by direct palpation or with the assistance of ultrasound without the need for interventional radiology
9. [Expansion] At least one injectable tumor (>=0.5cm in largest diameter) that can be injected either with or without the need for interventional radiology
10. [Expansion] Appropriate for treatment with either nivolumab or pembrolizumab
11. [Expansion] Progression following at least one prior regimen containing PD-1 directed immune checkpoint blockade
12. Measurable disease by RECIST v1.1
13. ECOG Performance Status of 0, 1, or 2
14. Resolution of any toxicity associated with prior therapy to ≤ Grade 1 (Residual toxicity of Grade 2 may be allowed following discussion with Medical Monitor)
15. Adequate hematologic function defined as:

    1. Absolute neutrophil count >=1,500/uL
    2. Platelet count >=100,000/uL
    3. [Expansion] Hemoglobin >=9 gm/dL
16. Adequate hepatic function defined as:

    1. Total bilirubin ≤ 1.5 x ULN
    2. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN

117. Adequate coagulation defined as:

1. International normalized ratio (INR) ≤ 1.5 x ULN or prothrombin time (PT) ≤ 1.5 x ULN
2. Partial thromboplastin time (PTT) or activated PTT (aPTT) ≤ 1.5 x ULN 18. Serum creatinine ≤ 1.5 x ULN or estimated GFR ≥ 60 mL/min/1.73 m2 (per MDRD GFR formula) 19. Women of childbearing potential must have a negative serum pregnancy test 20. All subjects of childbearing potential must be willing to consent to using effective contraception (as determined by the Investigator) while on treatment and for 3 months after their participation in the study ends

Exclusion Criteria:

1. Injectable tumor not sufficiently distanced from critical structures (e.g., major airway, neurovascular structure) where post injection swelling may place the subject at unacceptable risk
2. ≤ 21 days from prior anticancer therapy and C1D1 (e.g., chemotherapy, immunotherapy, intralesional therapy, irradiation therapy)
3. Known CNS metastases or leptomeningeal carcinomatosis, unless adequately treated and clinically stable off steroids for ≥ 14 days from C1D1
4. Severe infection requiring systemic antibiotic therapy or hospitalization for treatment of injection within 2 weeks of the first injection of VAX014
5. Need for systemic immunosuppressive therapy (≤10 mg of prednisone equivalent, or one time pulse steroids excepted)
6. Active autoimmune disease requiring systemic immunosuppressive therapy
7. No active lung disease or pneumonitis
8. No history of Grade 4 toxicity in response to prior PD-1 blockade
9. Any other malignancy likely to require treatment in the next 2 years (exceptions include cancer such as basal or squamous cell skin cancers, noninvasive cancer of the cervix, and local prostate cancer)
10. Known active infection with tuberculosis or HIV
11. Active Hepatitis B or C
12. [Females] pregnant or breastfeeding
13. Clinically significant cardiovascular abnormalities including:

    1. ≤ 12 months from prior MI
    2. Unstable angina pectoris
    3. ≤ 6 months from NYHA classification >3 CHF

10. Medical or psychological condition that places the subject at undue risk with study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of VAX014 | up to 21 days
  The MTD will be defined as the dose level at which at most one of six patients experiences a dose limiting toxicity (DLT) after 21 days of treatment have occurred, with the next higher dose having at least 2/3 or 2/6 patients experiencing a DLT
Incidence of Treatment-Emergency Adverse Events (Safety and Tolerability) | Through study completion, an average of 20 weeks
  Toxicities will be assessed in each subject by tracking the occurrence of graded Adverse Events (AEs). AEs will be graded according to the National Cancer Institute Common Terminology for Adverse Events (NCI CTCAE) v5.0
Recommended Phase 2 Dose (RP2D) for single agent intratumoral VAX014 | up to 5 weeks
  The RP2D will be determined following the determination of the MTD and with agreement by the Safety Review Committee
Acceptable dose of VAX014 in combination with PD-1 Inhibitor | 3 months
  Determine the acceptable dose of VAX014 when used in combination with Investigator's choice of nivolumab or pembrolizumab
Evaluation of efficacy of VAX014 in combination with either nivolumab or pembrolizumab | 18 months
  Evaluate efficacy including overall response rate (ORR), response of injected tumor(s) of VAX014 in combination with Investigator's choice of nivolumab or pembrolizumab

SECONDARY OUTCOMES:
Characterize systemic exposure by evaluating pharmacokinetics of intratumoral VAX014 as monotherapy and (if appropriate) in combination with nivolumab or pembrolizumab [systemic PK] | up to 1 week
  Whole blood will be collected for determination of VAX014 levels. PK data may demonstrate limited exposure or lack of detectable VAX014 in blood.
Anti-Drug Antibodies (Immunogenicity) [systemic ADA] | Up to 20 weeks
  The presence or absence of anti-drug antibodies (ADA) in serum will be assessed by assay in patients receiving VAX014 along or in combination with Investigator's choice of nivolumab or pembrolizumab
Overall Response Rate as VAX014 alone and in combination with either nivolumab or pembrolizumab | Up to 20 weeks
  Response rate will be evaluated for tumor lesions that will be assessed through CT, MRI, physical exam.

OTHER OUTCOMES:
Tumor Tissue (immune environment) | up to 8 weeks
  Tumor biopsies will be assessed for necrosis and immune changes within the tumor.
Anti-Tumor T Cells | Up to 20 weeks
  Changes in the number of Anti-Tumor T cells before and after treatment.
Cytokine levels | Up to 20 weeks
  Changes in the cytokine levels before and after treatment.
Type 1 IFN response | Up to 20 weeks
  Changes in type 1 IFN response before and after treatment.
STING expression | Baseline
  Predictive value of STING as a biomarker
RIG-I expression | Baseline
  Predictive value of RIG-I as a biomarker

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of Arizona Cancer Center, Tucson, Arizona
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - George Washington University, Washington D.C., District of Columbia
  - University of Maryland, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dartmouth Cancer Center, Lebanon, New Hampshire
  - Atlantic Health System, Morristown, New Jersey
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No